CLINICAL TRIAL: NCT02272010
Title: Targeted Alterations in n-3 and n-6 Fatty Acids for the Management of Mood Variability in the Maintenance Phase of Bipolar Disorder
Brief Title: Dietary Intervention for Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Erika Saunders, Associate Professor of Psychiatry, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Stanley-13T-013
Record Dates: First submitted 2014-08-18; First posted 2014-10-22 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental diet (Experimental): Altered n-6 and n-3 fatty acid intake.
  Interventions: Other: Experimental Diet
- Comparator Diet (Active Comparator): Diet standardized to usual n-6 and n-3 intake.
  Interventions: Other: Comparator Diet

INTERVENTIONS:
Other: Experimental Diet — Altered n-6 (linoleic acid) and n-3 (eicosapentaenic acid (EPA) + docosahexaenoic acid (DHA)) diet.
  Arms: Experimental diet
Other: Comparator Diet — Diet standardized to the usual American distribution of n-6 (7%) and n-3 EPA+DHA (150 mg per day).
  Arms: Comparator Diet

SUMMARY:
Bipolar disorder (BD) is a chronic, often disabling illness, and many individuals remain symptomatic despite pharmacotherapy. Significant mood variability often persists throughout the lifespan and predicts relapse, leading to functional impairment. Metabolism of dietary essential polyunsaturated fatty acids has been shown to be upstream of the neuroinflammatory processes that may lead to neurotoxicity and chronicity of illness in BD. The investigators hypothesize that an intervention diet designed to alter intake of polyunsaturated fatty acids that augments mood stabilizing medications will reduce inflammation; and that the reduction of inflammation will reduce mood variability in bipolar disorder. After a two-the investigatorsek baseline-monitoring period, the investigators will randomize individuals with BD to an intervention or a control diet. Mood will be measured daily using a smartphone. Phase 2 will consist of 12 the investigatorseks of a less intense intervention. Follow-up will then be completed at 6, 9, and 12 months post-baseline to assess for recurrence of mood episodes. By maintaining a certain diet in addition to taking mood-stabilizing medication, researchers hope to see whether specific dietary plans have any bearing on mood variability.

DETAILED DESCRIPTION:
The investigators will conduct a 2-arm, parallel group, randomized, controlled 24-week dietary intervention to evaluate the therapeutic efficacy of two dietary interventions in patients with BD. After a two-week baseline-monitoring period, the investigators will randomize 84 patients with chronic BD to augment usual treatment with either an experimentally-altered omega-3, omega-6 intervention or a control diet with average US intakes of n-3 and n-6 fatty acids. Subjects in both groups will remain under the care of their physician for the full duration of the trial. During the first phase of the trial (12 weeks), the intervention will be intense, during the second phase (12 weeks), a less intense intervention will be delivered, and after the two phases of intervention there will be a 24-week follow-up period.

The study is designed to achieve the following specific aims and obtain support for the following hypotheses:

Specific Aim 1 (primary mood outcome): To compare the efficacy of the experimental dietary intervention to the control diet in reducing variability of mood symptoms and reducing general psychological distress.

Hypothesis 1: Compared to the control diet, the experimental intervention will produce significant improvement in (1a) variability of daily mood symptoms, energy, and impulsivity using a Visual Analogue Scale measured using ecological momentary analysis (1); and (1b) psychological distress and general functioning using the PROMIS-29.

Specific Aim 2 (secondary mood outcome): To compare the efficacy of the experimental dietary intervention to the control diet in reducing recurrence.

Hypothesis 2: Compared to the control diet, the experimental intervention will produce significant reduction in recurrence of mood episodes over a 12-month period. To adequately power this study for measurement of recurrence, the investigators would need a sample size 2-3 times what the investigators estimate for this study, therefore the primary mood outcome is not recurrence of episode, but is measurement of mood variability, which in turn predicts recurrence. The investigators will measure recurrence to gather data for future studies.

Specific Aim 3 (primary biochemical outcome): To evaluate whether the experimental dietary intervention can alter n-6 AA and its bioactive metabolites, n-3 DHA and its bioactive metabolites in patients with BD.

Hypothesis 3: Compared to the control diet, the experimental intervention will significantly (1a) alter n-6 AA and n-3 DHA in erythrocytes; and (1b) alter 17-hydroxy DHA and reduce PGE2 in plasma.

Exploratory Aims: In an exploratory manner, the investigators will also (1) compare the efficacy of the experimental dietary intervention to the control diet in improving headache-related clinical endpoints in the subset of BP patients with comorbid migraines; (2) test the effects of the dietary interventions on a wide array of bioactive derivatives of n-3 and n-6 fatty acids and other inflammatory mediators (e.g. cytokines, CRP); and (3) evaluate whether biochemical alterations in n-3 DHA, n-6 AA and their bioactive metabolites are related to clinical improvements (4) compare the efficacy of the experimental dietary intervention to the control diet in preventing recurrence of illness in follow-up; (5) store samples for exploratory biomarker analysis.

ELIGIBILITY:
Inclusion Criteria:

1. BD - history of at least one manic or mixed episode
2. Clinically significant hypomania or depression
3. Current psychiatric treatment
4. Over 18

Exclusion Criteria:

1. Current hospitalization for BD
2. Active substance dependence or eating disorder
3. Active suicidal/homicidal ideation
4. Pregnancy
5. Active treatment for major medical illness
6. History of specific food allergies such as, but not limited to, fish, gluten, dairy products
7. Strong aversion to fish
8. Any condition or attitude which, in the opinion of the PI, would prevent full cooperation and commitment to the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2014-10; Primary Completion 2018-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Mood variability outcome | Measured from the 2-week baseline period to the 12-week period of the phase 1 intervention
  Each individual will be given a smartphone for fourteen weeks (2 weeks baseline plus 12 week phase 1 intervention) to measure facets of mood, sleep, and pain.

SECONDARY OUTCOMES:
Recurrence of mood episode | 1 year
  Recurrence will be measured through phone interviews and review of medical records.

OTHER OUTCOMES:
Plasma levels of omega-6 fatty acids | Comparing from baseline to weeks 4, 8, 12
  Group comparison of mean change from baseline in plasma levels of fatty acids, metabolites and lipidomics will be measured and analyzed in an exploratory fashion.
Psychological distress and general functioning | Baseline & weeks 0, 4, 8, 12
  Measured by PROMIS-29
Mood symptoms | Baseline & weeks 0, 4, 8, 12, 24, 48
  Mood, sleep, psychosocial stress and pain questionnaires.
Plasma levels of omega-3 fatty acids | Baseline & weeks 4, 8, 12
  Group comparison of mean change from baseline in plasma levels of fatty acids, metabolites and lipidomics will be measured and analyzed in an exploratory fashion.

CONTACTS AND LOCATIONS:
Overall Officials: Erika Saunders, M.D, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Milton S. Hershey Medical Center Clinical Research Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Bauer M, Glenn T, Alda M, Grof P, Sagduyu K, Bauer R, Lewitzka U, Whybrow PC. Comparison of pre-episode and pre-remission states using mood ratings from patients with bipolar disorder. Pharmacopsychiatry. 2011 May;44 Suppl 1:S49-53. doi: 10.1055/s-0031-1273765. Epub 2011 May 4. PMID 21544745
- [Background] Bauer M, Glenn T, Keil M, Bauer R, Marsh W, Grof P, Alda M, Sagduyu K, Murray G, Quiroz D, Baethge C, Whybrow PC. Brief depressive symptoms in patients with bipolar disorder: analysis of long-term self-reported data. Aust N Z J Psychiatry. 2012 Nov;46(11):1068-78. doi: 10.1177/0004867412452017. Epub 2012 Jun 25. PMID 22734088
- [Background] Bauer J, Gottfries GG, Forstl H. Critical comments on "Propionibacterium acnes in the cortex of patients with Alzheimer's disease" by H.H. Kornhuber (Eur Arch Psychiatry Clin Neurosci, 1996, 246:108-109). Eur Arch Psychiatry Clin Neurosci. 1996;246(4):224-6. doi: 10.1007/BF02188958. No abstract available. PMID 8832202
- [Background] aan het Rot M, Hogenelst K, Schoevers RA. Mood disorders in everyday life: a systematic review of experience sampling and ecological momentary assessment studies. Clin Psychol Rev. 2012 Aug;32(6):510-23. doi: 10.1016/j.cpr.2012.05.007. Epub 2012 Jun 6. PMID 22721999
- [Background] Jen A, Saunders EF, Ornstein RM, Kamali M, McInnis MG. Impulsivity, anxiety, and alcohol misuse in bipolar disorder comorbid with eating disorders. Int J Bipolar Disord. 2013 Aug 6;1:13. doi: 10.1186/2194-7511-1-13. eCollection 2013. PMID 25505680
- [Background] Bauer M, Glenn T, Whybrow PC, Grof P, Rasgon N, Alda M, Marsh W, Sagduyu K, Schmid R, Adli M. Changes in self-reported sleep duration predict mood changes in bipolar disorder. Psychol Med. 2008 Jul;38(7):1069-71. doi: 10.1017/S0033291708003280. Epub 2008 Apr 1. No abstract available. PMID 18377675
- [Background] Bauer M, Glenn T, Grof P, Pfennig A, Rasgon NL, Marsh W, Munoz RA, Sagduyu K, Alda M, Quiroz D, Sasse J, Whybrow PC. Self-reported data from patients with bipolar disorder: frequency of brief depression. J Affect Disord. 2007 Aug;101(1-3):227-33. doi: 10.1016/j.jad.2006.11.021. Epub 2007 Jan 16. PMID 17224186
- [Background] Myin-Germeys I, Oorschot M, Collip D, Lataster J, Delespaul P, van Os J. Experience sampling research in psychopathology: opening the black box of daily life. Psychol Med. 2009 Sep;39(9):1533-47. doi: 10.1017/S0033291708004947. Epub 2009 Feb 12. PMID 19215626
- [Background] Myin-Germeys I, Peeters F, Havermans R, Nicolson NA, DeVries MW, Delespaul P, Van Os J. Emotional reactivity to daily life stress in psychosis and affective disorder: an experience sampling study. Acta Psychiatr Scand. 2003 Feb;107(2):124-31. doi: 10.1034/j.1600-0447.2003.02025.x. PMID 12534438
- [Background] Keller MB, Lavori PW, Friedman B, Nielsen E, Endicott J, McDonald-Scott P, Andreasen NC. The Longitudinal Interval Follow-up Evaluation. A comprehensive method for assessing outcome in prospective longitudinal studies. Arch Gen Psychiatry. 1987 Jun;44(6):540-8. doi: 10.1001/archpsyc.1987.01800180050009. PMID 3579500
- [Background] Ramsden CE, Faurot KR, Zamora D, Suchindran CM, MacIntosh BA, Gaylord S, Ringel A, Hibbeln JR, Feldstein AE, Mori TA, Barden A, Lynch C, Coble R, Mas E, Palsson O, Barrow DA, Mann DJ. Targeted alteration of dietary n-3 and n-6 fatty acids for the treatment of chronic headaches: a randomized trial. Pain. 2013 Nov;154(11):2441-2451. doi: 10.1016/j.pain.2013.07.028. Epub 2013 Jul 22. PMID 23886520
- [Background] Merikangas KR, Akiskal HS, Angst J, Greenberg PE, Hirschfeld RM, Petukhova M, Kessler RC. Lifetime and 12-month prevalence of bipolar spectrum disorder in the National Comorbidity Survey replication. Arch Gen Psychiatry. 2007 May;64(5):543-52. doi: 10.1001/archpsyc.64.5.543. PMID 17485606
- [Background] Who. The World Health Report: 2001: Mental health: new understanding, new hope. Geneva: World Health Organization; 2001.
- [Background] Judd LL, Akiskal HS, Schettler PJ, Endicott J, Leon AC, Solomon DA, Coryell W, Maser JD, Keller MB. Psychosocial disability in the course of bipolar I and II disorders: a prospective, comparative, longitudinal study. Arch Gen Psychiatry. 2005 Dec;62(12):1322-30. doi: 10.1001/archpsyc.62.12.1322. PMID 16330720
- [Background] Judd LL, Akiskal HS, Schettler PJ, Endicott J, Maser J, Solomon DA, Leon AC, Rice JA, Keller MB. The long-term natural history of the weekly symptomatic status of bipolar I disorder. Arch Gen Psychiatry. 2002 Jun;59(6):530-7. doi: 10.1001/archpsyc.59.6.530. PMID 12044195
- [Background] Bauer M, Glenn T, Grof P, Schmid R, Pfennig A, Whybrow PC. Subsyndromal mood symptoms: a useful concept for maintenance studies of bipolar disorder? Psychopathology. 2010;43(1):1-7. doi: 10.1159/000255957. Epub 2009 Nov 6. PMID 19893338
- [Background] Kim HW, Rapoport SI, Rao JS. Altered arachidonic acid cascade enzymes in postmortem brain from bipolar disorder patients. Mol Psychiatry. 2011 Apr;16(4):419-28. doi: 10.1038/mp.2009.137. Epub 2009 Dec 29. PMID 20038946
- [Background] Rapoport SI, Basselin M, Kim HW, Rao JS. Bipolar disorder and mechanisms of action of mood stabilizers. Brain Res Rev. 2009 Oct;61(2):185-209. doi: 10.1016/j.brainresrev.2009.06.003. Epub 2009 Jun 23. PMID 19555719
- [Background] Berk M, Kapczinski F, Andreazza AC, Dean OM, Giorlando F, Maes M, Yucel M, Gama CS, Dodd S, Dean B, Magalhaes PV, Amminger P, McGorry P, Malhi GS. Pathways underlying neuroprogression in bipolar disorder: focus on inflammation, oxidative stress and neurotrophic factors. Neurosci Biobehav Rev. 2011 Jan;35(3):804-17. doi: 10.1016/j.neubiorev.2010.10.001. Epub 2010 Oct 8. PMID 20934453
- [Background] Reese EA, Cheon Y, Ramadan E, Kim HW, Chang L, Rao JS, Rapoport SI, Taha AY. Gabapentin's minimal action on markers of rat brain arachidonic acid metabolism agrees with its inefficacy against bipolar disorder. Prostaglandins Leukot Essent Fatty Acids. 2012 Aug-Sep;87(2-3):71-7. doi: 10.1016/j.plefa.2012.06.003. Epub 2012 Jul 27. PMID 22841517
- [Background] Cheon Y, Park JY, Modi HR, Kim HW, Lee HJ, Chang L, Rao JS, Rapoport SI. Chronic olanzapine treatment decreases arachidonic acid turnover and prostaglandin E(2) concentration in rat brain. J Neurochem. 2011 Oct;119(2):364-76. doi: 10.1111/j.1471-4159.2011.07410.x. Epub 2011 Sep 20. PMID 21812779
- [Background] Rao JS, Harry GJ, Rapoport SI, Kim HW. Increased excitotoxicity and neuroinflammatory markers in postmortem frontal cortex from bipolar disorder patients. Mol Psychiatry. 2010 Apr;15(4):384-92. doi: 10.1038/mp.2009.47. Epub 2009 Jun 2. PMID 19488045
- [Background] Rao JS, Keleshian VL, Klein S, Rapoport SI. Epigenetic modifications in frontal cortex from Alzheimer's disease and bipolar disorder patients. Transl Psychiatry. 2012 Jul 3;2(7):e132. doi: 10.1038/tp.2012.55. PMID 22760556
- [Background] Hibbeln JR, Palmer JW, Davis JM. Are disturbances in lipid-protein interactions by phospholipase-A2 a predisposing factor in affective illness? Biol Psychiatry. 1989 Apr 1;25(7):945-61. doi: 10.1016/0006-3223(89)90274-6. PMID 2566335
- [Background] Chiu CC, Huang SY, Su KP, Lu ML, Huang MC, Chen CC, Shen WW. Polyunsaturated fatty acid deficit in patients with bipolar mania. Eur Neuropsychopharmacol. 2003 Mar;13(2):99-103. doi: 10.1016/s0924-977x(02)00130-x. PMID 12650953
- [Background] Sublette ME, Bosetti F, DeMar JC, Ma K, Bell JM, Fagin-Jones S, Russ MJ, Rapoport SI. Plasma free polyunsaturated fatty acid levels are associated with symptom severity in acute mania. Bipolar Disord. 2007 Nov;9(7):759-65. doi: 10.1111/j.1399-5618.2007.00387.x. PMID 17988367
- [Background] McNamara RK, Jandacek R, Rider T, Tso P, Dwivedi Y, Pandey GN. Selective deficits in erythrocyte docosahexaenoic acid composition in adult patients with bipolar disorder and major depressive disorder. J Affect Disord. 2010 Oct;126(1-2):303-11. doi: 10.1016/j.jad.2010.03.015. Epub 2010 Apr 21. PMID 20413162
- [Background] Evans SJ, Prossin AR, Harrington GJ, Kamali M, Ellingrod VL, Burant CF, McInnis MG. Fats and factors: lipid profiles associate with personality factors and suicidal history in bipolar subjects. PLoS One. 2012;7(1):e29297. doi: 10.1371/journal.pone.0029297. Epub 2012 Jan 13. PMID 22253709
- [Background] Evans SJ, Kamali M, Prossin AR, Harrington GJ, Ellingrod VL, McInnis MG, Burant CF. Association of plasma omega-3 and omega-6 lipids with burden of disease measures in bipolar subjects. J Psychiatr Res. 2012 Nov;46(11):1435-41. doi: 10.1016/j.jpsychires.2012.07.016. Epub 2012 Aug 11. PMID 22884424
- [Background] Basselin M, Kim HW, Chen M, Ma K, Rapoport SI, Murphy RC, Farias SE. Lithium modifies brain arachidonic and docosahexaenoic metabolism in rat lipopolysaccharide model of neuroinflammation. J Lipid Res. 2010 May;51(5):1049-56. doi: 10.1194/jlr.M002469. Epub 2009 Dec 29. PMID 20040630 (Retraction: PMID 30068753 J Lipid Res. 2018 Aug;59(8):1547)
- [Background] Antonova M, Wienecke T, Olesen J, Ashina M. Prostaglandin E(2) induces immediate migraine-like attack in migraine patients without aura. Cephalalgia. 2012 Aug;32(11):822-33. doi: 10.1177/0333102412451360. Epub 2012 Jun 19. PMID 22718556
- [Background] Soares JK, Rocha-de-Melo AP, Medeiros MC, Queiroga RC, Bomfim MA, de Souza AF, Nascimento AL, Guedes RC. Conjugated linoleic acid in the maternal diet differentially enhances growth and cortical spreading depression in the rat progeny. Biochim Biophys Acta. 2012 Oct;1820(10):1490-5. doi: 10.1016/j.bbagen.2012.05.010. Epub 2012 Jun 1. PMID 22659523
- [Background] BALANCE investigators and collaborators; Geddes JR, Goodwin GM, Rendell J, Azorin JM, Cipriani A, Ostacher MJ, Morriss R, Alder N, Juszczak E. Lithium plus valproate combination therapy versus monotherapy for relapse prevention in bipolar I disorder (BALANCE): a randomised open-label trial. Lancet. 2010 Jan 30;375(9712):385-95. doi: 10.1016/S0140-6736(09)61828-6. Epub 2010 Jan 19. PMID 20092882
- [Background] Linde M, Mulleners WM, Chronicle EP, McCrory DC. Valproate (valproic acid or sodium valproate or a combination of the two) for the prophylaxis of episodic migraine in adults. Cochrane Database Syst Rev. 2013 Jun 24;2013(6):CD010611. doi: 10.1002/14651858.CD010611. PMID 23797677
- [Background] Noaghiul S, Hibbeln JR. Cross-national comparisons of seafood consumption and rates of bipolar disorders. Am J Psychiatry. 2003 Dec;160(12):2222-7. doi: 10.1176/appi.ajp.160.12.2222. PMID 14638594
- [Background] Hibbeln JR, Nieminen LR, Blasbalg TL, Riggs JA, Lands WE. Healthy intakes of n-3 and n-6 fatty acids: estimations considering worldwide diversity. Am J Clin Nutr. 2006 Jun;83(6 Suppl):1483S-1493S. doi: 10.1093/ajcn/83.6.1483S. PMID 16841858
- [Background] Freeman MP, Hibbeln JR, Wisner KL, Davis JM, Mischoulon D, Peet M, Keck PE Jr, Marangell LB, Richardson AJ, Lake J, Stoll AL. Omega-3 fatty acids: evidence basis for treatment and future research in psychiatry. J Clin Psychiatry. 2006 Dec;67(12):1954-67. doi: 10.4088/jcp.v67n1217. PMID 17194275
- [Background] Kraguljac NV, Montori VM, Pavuluri M, Chai HS, Wilson BS, Unal SS. Efficacy of omega-3 fatty acids in mood disorders - a systematic review and metaanalysis. Psychopharmacol Bull. 2009;42(3):39-54. PMID 19752840
- [Background] Stoll AL, Locke CA, Marangell LB, Severus WE. Omega-3 fatty acids and bipolar disorder: a review. Prostaglandins Leukot Essent Fatty Acids. 1999 May-Jun;60(5-6):329-37. doi: 10.1016/s0952-3278(99)80008-8. PMID 10471117
- [Background] Stoll AL, Severus WE, Freeman MP, Rueter S, Zboyan HA, Diamond E, Cress KK, Marangell LB. Omega 3 fatty acids in bipolar disorder: a preliminary double-blind, placebo-controlled trial. Arch Gen Psychiatry. 1999 May;56(5):407-12. doi: 10.1001/archpsyc.56.5.407. PMID 10232294
- [Background] Keck PE Jr, Mintz J, McElroy SL, Freeman MP, Suppes T, Frye MA, Altshuler LL, Kupka R, Nolen WA, Leverich GS, Denicoff KD, Grunze H, Duan N, Post RM. Double-blind, randomized, placebo-controlled trials of ethyl-eicosapentanoate in the treatment of bipolar depression and rapid cycling bipolar disorder. Biol Psychiatry. 2006 Nov 1;60(9):1020-2. doi: 10.1016/j.biopsych.2006.03.056. Epub 2006 Jun 30. PMID 16814257
- [Background] Murphy BL, Stoll AL, Harris PQ, Ravichandran C, Babb SM, Carlezon WA Jr, Cohen BM. Omega-3 fatty acid treatment, with or without cytidine, fails to show therapeutic properties in bipolar disorder: a double-blind, randomized add-on clinical trial. J Clin Psychopharmacol. 2012 Oct;32(5):699-703. doi: 10.1097/JCP.0b013e318266854c. PMID 22926607
- [Background] Frangou S, Lewis M, McCrone P. Efficacy of ethyl-eicosapentaenoic acid in bipolar depression: randomised double-blind placebo-controlled study. Br J Psychiatry. 2006 Jan;188:46-50. doi: 10.1192/bjp.188.1.46. PMID 16388069
- [Background] Frangou S, Lewis M, Wollard J, Simmons A. Preliminary in vivo evidence of increased N-acetyl-aspartate following eicosapentanoic acid treatment in patients with bipolar disorder. J Psychopharmacol. 2007 Jun;21(4):435-9. doi: 10.1177/0269881106067787. Epub 2006 Aug 4. PMID 16891338
- [Background] Rao JS, Kim HW, Kellom M, Greenstein D, Chen M, Kraft AD, Harry GJ, Rapoport SI, Basselin M. Increased neuroinflammatory and arachidonic acid cascade markers, and reduced synaptic proteins, in brain of HIV-1 transgenic rats. J Neuroinflammation. 2011 Aug 16;8:101. doi: 10.1186/1742-2094-8-101. PMID 21846384 (Retraction: PMID 28482852 J Neuroinflammation. 2017 May 9;14 (1):95)
- [Background] Kim HW, Rapoport SI, Rao JS. Altered expression of apoptotic factors and synaptic markers in postmortem brain from bipolar disorder patients. Neurobiol Dis. 2010 Mar;37(3):596-603. doi: 10.1016/j.nbd.2009.11.010. Epub 2009 Nov 26. PMID 19945534
- [Background] Rapoport SI. Arachidonic acid and the brain. J Nutr. 2008 Dec;138(12):2515-20. doi: 10.1093/jn/138.12.2515. PMID 19022981
- [Background] Modi HR, Taha AY, Kim HW, Chang L, Rapoport SI, Cheon Y. Chronic clozapine reduces rat brain arachidonic acid metabolism by reducing plasma arachidonic acid availability. J Neurochem. 2013 Feb;124(3):376-87. doi: 10.1111/jnc.12078. Epub 2012 Dec 6. PMID 23121637
- [Background] Kim HW, Cheon Y, Modi HR, Rapoport SI, Rao JS. Effects of chronic clozapine administration on markers of arachidonic acid cascade and synaptic integrity in rat brain. Psychopharmacology (Berl). 2012 Aug;222(4):663-74. doi: 10.1007/s00213-012-2671-7. Epub 2012 Mar 14. PMID 22414961
- [Background] Shimshoni JA, Basselin M, Li LO, Coleman RA, Rapoport SI, Modi HR. Valproate uncompetitively inhibits arachidonic acid acylation by rat acyl-CoA synthetase 4: relevance to valproate's efficacy against bipolar disorder. Biochim Biophys Acta. 2011 Mar;1811(3):163-9. doi: 10.1016/j.bbalip.2010.12.006. Epub 2010 Dec 22. PMID 21184843
- [Background] Lee HJ, Rao JS, Chang L, Rapoport SI, Kim HW. Chronic imipramine but not bupropion increases arachidonic acid signaling in rat brain: is this related to 'switching' in bipolar disorder? Mol Psychiatry. 2010 Jun;15(6):602-14. doi: 10.1038/mp.2008.117. Epub 2008 Nov 4. PMID 18982003
- [Background] Rao JS, Rapoport SI. Mood-stabilizers target the brain arachidonic acid cascade. Curr Mol Pharmacol. 2009 Jun;2(2):207-14. doi: 10.2174/1874467210902020207. PMID 20021459
- [Background] Lee HJ, Ertley RN, Rapoport SI, Bazinet RP, Rao JS. Chronic administration of lamotrigine downregulates COX-2 mRNA and protein in rat frontal cortex. Neurochem Res. 2008 May;33(5):861-6. doi: 10.1007/s11064-007-9526-3. Epub 2007 Dec 14. PMID 18080190
- [Background] Vieta E. Guide to Assessment Scales in Bipolar Disorder. 2 ed. London, UK: Current Medicine Group Ltd; 2010.
- [Background] Snaith RP, Harrop FM, Newby DA, Teale C. Grade scores of the Montgomery-Asberg Depression and the Clinical Anxiety Scales. Br J Psychiatry. 1986 May;148:599-601. doi: 10.1192/bjp.148.5.599. No abstract available. PMID 3779233
- [Background] Ruissen AM, Widdershoven GA, Meynen G, Abma TA, van Balkom AJ. A systematic review of the literature about competence and poor insight. Acta Psychiatr Scand. 2012 Feb;125(2):103-13. doi: 10.1111/j.1600-0447.2011.01760.x. Epub 2011 Sep 8. PMID 21902676
- [Background] Bauer M, Wilson T, Neuhaus K, Sasse J, Pfennig A, Lewitzka U, Grof P, Glenn T, Rasgon N, Bschor T, Whybrow PC. Self-reporting software for bipolar disorder: validation of ChronoRecord by patients with mania. Psychiatry Res. 2008 Jun 30;159(3):359-66. doi: 10.1016/j.psychres.2007.04.013. Epub 2008 Apr 18. PMID 18423616
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Davidson J, Turnbull CD, Strickland R, Miller R, Graves K. The Montgomery-Asberg Depression Scale: reliability and validity. Acta Psychiatr Scand. 1986 May;73(5):544-8. doi: 10.1111/j.1600-0447.1986.tb02723.x. PMID 3751660
- [Background] Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry. 1979 Apr;134:382-9. doi: 10.1192/bjp.134.4.382. PMID 444788
- [Background] Altman EG, Hedeker DR, Janicak PG, Peterson JL, Davis JM. The Clinician-Administered Rating Scale for Mania (CARS-M): development, reliability, and validity. Biol Psychiatry. 1994 Jul 15;36(2):124-34. doi: 10.1016/0006-3223(94)91193-2. PMID 7948445
- [Background] Young RC, Biggs JT, Ziegler VE, Meyer DA. A rating scale for mania: reliability, validity and sensitivity. Br J Psychiatry. 1978 Nov;133:429-35. doi: 10.1192/bjp.133.5.429. PMID 728692
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Horne JA, Ostberg O. A self-assessment questionnaire to determine morningness-eveningness in human circadian rhythms. Int J Chronobiol. 1976;4(2):97-110. PMID 1027738
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Gray MJ, Litz BT, Hsu JL, Lombardo TW. Psychometric properties of the life events checklist. Assessment. 2004 Dec;11(4):330-41. doi: 10.1177/1073191104269954. PMID 15486169
- [Background] Vinokur AD, van Ryn M. Social support and undermining in close relationships: their independent effects on the mental health of unemployed persons. J Pers Soc Psychol. 1993 Aug;65(2):350-9. doi: 10.1037//0022-3514.65.2.350. PMID 8366424
- [Background] McKee SA AM, Kochetkova A, Maciejewski P, O'Malley S, Krishnan-Sarin S, & Mazure CM. A new measure for assessing the impact of stressful events on smoking behavior. Annual Meeting of the Society for Research on Nicotine and Tobacco; Prague, CZ2005. p. 16.
- [Background] Saunders JB, Aasland OG, Babor TF, de la Fuente JR, Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. Addiction. 1993 Jun;88(6):791-804. doi: 10.1111/j.1360-0443.1993.tb02093.x. PMID 8329970
- [Background] Stewart WF, Lipton RB, Kolodner KB, Sawyer J, Lee C, Liberman JN. Validity of the Migraine Disability Assessment (MIDAS) score in comparison to a diary-based measure in a population sample of migraine sufferers. Pain. 2000 Oct;88(1):41-52. doi: 10.1016/S0304-3959(00)00305-5. PMID 11098098
- [Background] Stewart WF, Lipton RB, Whyte J, Dowson A, Kolodner K, Liberman JN, Sawyer J. An international study to assess reliability of the Migraine Disability Assessment (MIDAS) score. Neurology. 1999 Sep 22;53(5):988-94. doi: 10.1212/wnl.53.5.988. PMID 10496257
- [Background] Kosinski M, Bayliss MS, Bjorner JB, Ware JE Jr, Garber WH, Batenhorst A, Cady R, Dahlof CG, Dowson A, Tepper S. A six-item short-form survey for measuring headache impact: the HIT-6. Qual Life Res. 2003 Dec;12(8):963-74. doi: 10.1023/a:1026119331193. PMID 14651415
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Siddiqui O, Hung HM, O'Neill R. MMRM vs. LOCF: a comprehensive comparison based on simulation study and 25 NDA datasets. J Biopharm Stat. 2009;19(2):227-46. doi: 10.1080/10543400802609797. PMID 19212876
- [Background] Hamer RM, Simpson PM. Last observation carried forward versus mixed models in the analysis of psychiatric clinical trials. Am J Psychiatry. 2009 Jun;166(6):639-41. doi: 10.1176/appi.ajp.2009.09040458. No abstract available. PMID 19487398
- [Derived] Saunders EFH, Mukherjee D, Myers T, Wasserman E, Hameed A, Bassappa Krishnamurthy V, MacIntosh B, Domenichiello A, Ramsden CE, Wang M. Adjunctive dietary intervention for bipolar disorder: a randomized, controlled, parallel-group, modified double-blinded trial of a high n-3 plus low n-6 diet. Bipolar Disord. 2022 Mar;24(2):171-184. doi: 10.1111/bdi.13112. Epub 2021 Aug 2. PMID 34218509
- [Derived] Huesch MD, Mukherjee D, Saunders EF. E-recruitment into a bipolar disorder trial using Facebook tailored advertising. Clin Trials. 2018 Oct;15(5):522-523. doi: 10.1177/1740774518784018. Epub 2018 Jun 28. No abstract available. PMID 29952243